CLINICAL TRIAL: NCT00868179
Title: A Cohort (Follow Up) Study With 100 Subjects Having a Primary Total Knee Replacement, Taking Pradax (Tablet) Post Discharge for Ten Days, Without the Need for Routine Coagulation Monitoring and Dose Adjustment
Brief Title: A Cohort Study With 100 Subjects Having a Primary Total Knee Replacement, Taking Pradax Post Discharge for Ten Days
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study never started
Sponsor: Ross Leighton (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Ross Leighton, Orthopedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pradax
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Thromboembolism
Keywords: Thrombosis; total knee replacement
MeSH Terms: conditions — Thromboembolism; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pradax (Experimental): This is the only arm in the study and all will follow the same protocol for the study which is taking the pradax after total knee replacement
  Interventions: Drug: Pradax

INTERVENTIONS:
Drug: Pradax — Pradax (dabigatran etexilate) is a prodrug that when converted to the active from in the liver and plasma it becomes a reversible, competitive direct thrombin inhibitor. Thrombin catalyses the conversion of soluble fibrinogen into soluble fibrin, the final step in the coagulation cascade. Pradax competitively blocks the active site of both free and clot-bound thrombin, preventing the development of a thrombus. they will take 110 mg 1-4 hours post op. and 220mg daily until 10 days post op.
  Other Names: Pradax dabigatran etexilate

SUMMARY:
Currently standard of care for preventing blood clots in total knee replacement patients is the drug Fragmin which is a daily injection for 10 days after surgery. Patients are in hospital for 3 to 5 days after total knee replacement surgery and patients are taught in hospital to do their injections.

The investigators would like to introduce the drug Pradax. Pradax is a Health Canada approved once a day, oral drug that may prevent blood clots in the patient's leg. In this study the patient will receive the standard of care injection drug Fragmin while in hospital but on discharge home the patient will take the oral drug Pradax daily (2 tablets 110mg) for 10 days.

DETAILED DESCRIPTION:
We will enroll one hundred patients who are scheduled to have a total knee replacement. If you have signed the consent form for this study you will receive the standard of care treatment for blood clots, which is a daily injection drug called Fragmin. On the day of discharge from hospital study patients will receive a ten day supply of oral Pradax. to be taken once a day. The Orthopaedic research coordinator will call the study patients at post discharge day three and five to check on compliance and or concerns. All total knee replacement patients whether in study or not are seen in the Orthopaedic clinic at post op day 10 for staple removal and again at the 6 week point, 3 month, and 6 month and 1 year point. Standard of care x-rays are done also at these visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for the study if they are adult age, being greater than 18 years of age and less than 95 years of age. They must have the indications for a total knee replacement and have sufficiently passed the medically necessary tests by their surgeon to warrant total knee replacement.

Exclusion Criteria:

* Patients with active bleeding, or high risk of bleeding that contra-indicates the use of Pradax
* Renal or liver contra-indication necessitating adjustments of its dose.
* Clinically significant liver disease,
* Concomitant use of Proteus Ace inhibitors
* The use of the human immunitive deficiency virus
* The use of fibrinolynic agents
* Planned intermittent pneumatic compression or requirement of ongoing anticoagulation therapy
* Pregnancy
* Breast-feeding.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy outcome will be the clinical evidence of any deep vein thrombosis, non-fatal pulmonary embolism or death from any causes within 28 days after surgery. The primary safety outcome is major bleeding | 28 day post op and 6 months radiograophically

SECONDARY OUTCOMES:
Secondary efficacy end points will be the radiographic assessment of healing, the clinical assessment of weight-¬bearing status at 6 months post treatment, and the incidence of additional surgical/medical interventions to promote healing. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ross K Leighton, MD FRCSC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada